CLINICAL TRIAL: NCT01727050
Title: Randomized Prospective Trial of Fibrin Sealant Spray Versus Mechanical Stapling in Laparoscopic Totally Extraperitoneal Hernioplasty
Brief Title: Fibrin Sealant Spray Versus Mechanical Stapling in Laparoscopic Totally Extraperitoneal Hernioplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anthony Teoh, Honorary Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FSMSLH
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mechanical stapling (Active Comparator)
  Interventions: Device: Mechanical stapling
- Fibrin sealant spray (Active Comparator)
  Interventions: Device: Fibrin sealant spray

INTERVENTIONS:
Device: Fibrin sealant spray — Fixation of mesh would be performed using fibrin sealant spray applied with a laparoscopic spray catheter
  Arms: Fibrin sealant spray
Device: Mechanical stapling — Fixation of mesh would be performed using mechanical staplers
  Arms: Mechanical stapling

SUMMARY:
Laparoscopic totally extraperitoneal hernioplasty (TEP) is one of the treatment options for the repair of primary unilateral inguinal hernia. Previous studies showed that patients underwent TEP have less post-operative pain and earlier return to normal activities. However, chronic pain is still a major issue affecting quality of life after TEP with a reported incidence of 9.2-22.5%. Mechanical stapling is the most commonly used method of mesh fixation to prevent mesh migration but nerve entrapment by staples causing intractable pain had been reported. Recently several clinical trials showed that mesh fixation with fibrin sealant (FS) in TEP resulted in less chronic pain but increased incidence of seroma. A spraying device for application of FS laparoscopically is now available which can achieve mesh fixation by using fewer amounts of FS.

In this study, the investigators aim to compare the effectiveness of using fibrin spray for mesh fixation in reducing chronic pain after TEP. The investigators performed a randomized controlled trial by allocating patients in two study arm in random manner. The treatment group will have the mesh fixed by fibrin sealant spray, whereas the control group will have conventional mechanical staples for fixation. Operative procedures and post-operative management for the 2 groups will be identical. They will be follow-up at 1-month and 6-month after operation to evaluate the operative results and the incidence of chronic pain. Any complications related to the mesh and operation will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive male patients aged between 18 to 70 years with reducible unilateral inguinal hernia undergoing day-case TEP under general anaesthesia will be considered eligible.

Exclusion Criteria:

* Bilateral hernia, recurrent hernia, partially reducible or strangulated hernia, large inguinal-scrotal hernia, previous abdominal incision (including previous contralateral hernia repair), peripheral neuropathy, coagulopathy or taking anticoagulation drugs, end-stage renal failure, cirrhosis, impaired cognitive function and those not consent to study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2007-06; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence of chronic pain | 6 months

SECONDARY OUTCOMES:
Severity of acute pain | 1 week
Morbidities | 30 day
Recurrence rate | 6 month
Quality of life assessment | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Chan MS, Teoh AY, Chan KW, Tang YC, Ng EK, Leong HT. Randomized double-blinded prospective trial of fibrin sealant spray versus mechanical stapling in laparoscopic total extraperitoneal hernioplasty. Ann Surg. 2014 Mar;259(3):432-7. doi: 10.1097/SLA.0b013e3182a6c513. PMID 24045438